CLINICAL TRIAL: NCT01521546
Title: Early Treatment With Aldosterone Antagonism Attenuates Cardiomyopathy in Duchenne Muscular Dystrophy
Brief Title: Eplerenone for Subclinical Cardiomyopathy in Duchenne Muscular Dystrophy
Acronym: E-SCAR DMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Subha Raman (Other)
Collaborators: Ballou Skies (Other)
Responsible Party: Sponsor-Investigator, Subha Raman, Professor of Medicine, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011H0251
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; cardiomyopathy; aldosterone antagonist
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Cardiomyopathies | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eplerenone (Active Comparator): active study drug
  Interventions: Drug: eplerenone
- sugar pill (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: eplerenone — 25mg tablet, once daily by mouth for 12 months
  Arms: eplerenone
Drug: placebo — one tablet by mouth daily for 12 months
  Arms: sugar pill

SUMMARY:
Duchenne muscular dystrophy (DMD), the most common muscular dystrophy, leads to skeletal and cardiac muscle damage. Treatment of pulmonary complications has improved survival; however, heart muscle disease or cardiomyopathy has emerged as a leading cause of death, typically by the third decade. Although myocardial changes begin early, clinically significant heart disease is rarely detected in the first decade of life. Consequently, DMD cardiomyopathy frequently goes unrecognized (and untreated) until advanced (and irreversible).

Current DMD cardiovascular care guidelines recommend beta-blockers and angiotensin converting enzyme inhibitors (ACEIs) when decreased ejection fraction (EF) is noted by echocardiography (echo); however, this strategy has not significantly improved outcomes. Our team has recently made a breakthrough in a mouse study, showing in a model that causes the same heart muscle disease in humans with DMD adding an old medicine traditionally used for high blood pressure and late-stage heart failure can actually prevent heart muscle damage. Because of this drug's proven safety in both children and adults, it is ready to be studied immediately in an RCT in patients with DMD to hopefully show, as we did in mice, that we can prevent the devastating consequences of heart muscle damage.

DETAILED DESCRIPTION:
Duchenne Muscular dystrophy (DMD) is a deadly X-linked disease affecting 1 in 3,500 males. DMD patients suffer significant disability due to skeletal myopathy and excess death due to cardiomyopathy. Current guidelines advocate initiating cardioprotective treatment with evident global cardiac dysfunction, yet this treatment paradigm has not improved survival much beyond the third decade of life. Potentially promising approaches like gene therapy will take considerable time to improve outcomes. Recently completed studies in a DMD mouse model at our institution indicate that existing drugs known as aldosterone antagonists, typically reserved for advanced heart failure patients, preserve skeletal and cardiac muscle function at 80% of normal. Clinical studies at many centers including ours have shown that high-resolution, noninvasive cardiac magnetic resonance (CMR) detects subclinical myocardial fibrosis and abnormal regional function prior to global functional abnormalities. Combining findings from these preclinical and clinical studies, we plan to execute a randomized, controlled clinical trial (RCT) of eplerenone plus background therapy vs. background therapy alone in patients with DMD. We expect that the aldosterone antagonist eplerenone compared to standard therapy significantly delays progressive cardiomyopathy and skeletal myopathy using highly reproducible imaging biomarkers selected for efficient sample size design, to ultimately reduce disability and death.

ELIGIBILITY:
Inclusion Criteria:

* DMD patients age 7 years and older (and able to complete cardiac MRI without sedation) with preserved left ventricular (LV) systolic function and abnormal heart muscle by late post-gadolinium imaging (LGE)

Exclusion Criteria:

* renal insufficiency (GFR <40 mL/min/m2)
* non-MR compatible implants (e.g. neurostimulator, AICD)
* severe claustrophobia
* allergy to gadolinium contrast
* prior use of or known allergy to epleronone
* use of potassium-sparing diuretics
* serum potassium level of >5.0 mmol/L

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subha V Raman, MD, MSEE, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Mattel Children's Hospital and David Geffen School of Medicine at UCLA, Los Angeles, California
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Derived] Raman SV, Hor KN, Mazur W, He X, Kissel JT, Smart S, McCarthy B, Roble SL, Cripe LH. Eplerenone for early cardiomyopathy in Duchenne muscular dystrophy: results of a two-year open-label extension trial. Orphanet J Rare Dis. 2017 Feb 20;12(1):39. doi: 10.1186/s13023-017-0590-8. PMID 28219442
- [Derived] Raman SV, Hor KN, Mazur W, Halnon NJ, Kissel JT, He X, Tran T, Smart S, McCarthy B, Taylor MD, Jefferies JL, Rafael-Fortney JA, Lowe J, Roble SL, Cripe LH. Eplerenone for early cardiomyopathy in Duchenne muscular dystrophy: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2015 Feb;14(2):153-61. doi: 10.1016/S1474-4422(14)70318-7. Epub 2014 Dec 30. PMID 25554404

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was required prior to assignment.
Groups:
- Placebo: placebo
  placebo: one tablet by mouth daily for 12 months
Period: Overall Study
Arm/Group | Placebo | Eplerenone
Started | 22 | 20
Completed | 20 | 20
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Males with Duchenne Muscular Dystrophy
Groups:
- Total: Total of all reporting groups
Arm/Group | Eplerenone | Placebo | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Age | 14.5 [12.0 to 18.5] | 15.0 [11.0 to 19.0] | 15.0 [11.75 to 19.0]
Sex: Female, Male [Count of Participants; unit: Participants] — The study was approved for 42 participants and 42 participants were enrolled.
  Participants
    Female | 0 | 0 | 0
    Male | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: 12-month Change in Myocardial Strain
Description: a sensitive measurement of heart function using cardiac MRI, change was 12 months minus baseline.
Time Frame: baseline and 12 months
Measure: Median (Inter-Quartile Range); unit: percent change in heart dimension
Groups:
- Eplerenone: eplerenone one tablet by mouth daily for 12 months
Arm/Group | Placebo | Eplerenone
Number analyzed (Participants) | 20 | 20
percent change in heart dimension | 2.2 [1.3 to 3.1] | 1.0 [0.3 to 2.2]

ADVERSE EVENTS:
Groups:
- Placebo: placebo one tablet daily for 12 months
- Eplerenone: eplerenone one tablet daily for 12 months
Arm/Group | Placebo | Eplerenone
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/20
Other Adverse Events (participants affected / at risk) | 2/22 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | Eplerenone (N=20)
death due to fat embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | Eplerenone (N=20)
flushing (Skin and subcutaneous tissue disorders) | 1 | 0
anxiety (Psychiatric disorders) | 1 | 0
headache coincident with seasonal allergies (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No